CLINICAL TRIAL: NCT07058337
Title: Methotrexate as an Adjunct to Parsplana Vitrectomy for the Preventing and Treatment of Proliferative Vitreoretinopathy in Rhegmatogenous Retinal Detachment: A Clinical Study
Brief Title: Methotrexate in Retinal Detachment With Proliferative Vitreoretinopathy
Acronym: Methotrexate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Methorexate in PVR
Record Dates: First submitted 2025-04-28; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Retinal Detachment
Keywords: Proliferative Vitreoretinopathy; Rhegmatogenous Retinal Detachment; Methotrexate
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (PPV Alone) (Active Comparator): Patients in this group will undergo pars plana vitrectomy (PPV) only.
  Interventions: Procedure: parsplana vitrectomy
- Group 2 (PPV with Methotrexate) (Active Comparator): Patients in this group will receive complete PPV along with adjunctive intravitreal methotrexate
  Interventions: Procedure: parsplana vitrectomy; Procedure: adjunctive use of Methotrexate

INTERVENTIONS:
Procedure: parsplana vitrectomy — 23 gauge parsplana vitrectomy
Procedure: adjunctive use of Methotrexate — intravitreal methotrexate (200 μg/0.05 ml) at the time of surgery and repeated weekly for four weeks postoperatively
  Arms: Group 2 (PPV with Methotrexate)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intraocular methotrexate (MTX) in preventing and managing proliferative vitreoretinopathy (PVR) in patients undergoing retinal detachment surgery

DETAILED DESCRIPTION:
Patients will be randomized into two groups if clinical evidence of PVR is detected at the time of surgery, utilizing a computer-generated list for randomization. All surgeries will be conducted by the same surgeon to maintain consistency in technique.

Intervention Groups:

1. Group 1 (PPV Alone): Patients in this group will undergo pars plana vitrectomy (PPV) only.

Group 2 (PPV with Methotrexate): Patients in this group will receive complete PPV along with adjunctive intravitreal methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Diagnosed with RRD with clinical signs of PVR.
* No history of prior ocular surgeries for RRD or PVR.

Exclusion Criteria:

* Patients with other retinal diseases (e.g., diabetic retinopathy or retinal vascular occlusions).
* Individuals with significant systemic illnesses that could influence surgical outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 and 6 months after tamponade removal
  Best-Corrected Visual Acuity (BCVA):
  BCVA will be measured using the logarithm of the minimum angle of resolution (LogMAR) scale. A LogMAR value of 0.0 corresponds to normal visual acuity (Snellen equivalent 6/6 or 20/20), representing the ability to resolve an optotype that subtends 5 minutes of arc. Visual acuity will be converted to LogMAR values for statistical analysis.
Anatomical Success | within 6 months after tamponade removal
  Successful Retinal Reattachment:
  Defined as complete reattachment of the neurosensory retina to the underlying retinal pigment epithelium (RPE) without persistent or recurrent subretinal fluid at the final follow-up visit, as confirmed by clinical examination and optical coherence tomography (OCT), in the absence of tamponade or additional surgical intervention.
Number of Operations Required | within 6 months after tamponade removal
  The total number of surgical procedures (including vitrectomy, scleral buckling, retinopexy, or tamponade exchange) required to achieve and maintain retinal reattachment will be recorded for each eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebsar Eye Center, Cairo, Egypt, Egypt